CLINICAL TRIAL: NCT03311282
Title: Evaluation of the New Chicco Breast-like and Evolutive Feeding Bottles on Physiological Feeding Parameters and Colic-like Symptoms in Infants
Brief Title: New Chicco Bottles Study
Acronym: Step-Up
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sprim Advanced Life Sciences (Other)
Collaborators: Artsana S.p.a. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Art001
Record Dates: First submitted 2017-10-04; First posted 2017-10-17 (Actual); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Feeding Behavior
Keywords: breastfeeding; infants; squeezing; breathing
MeSH Terms: conditions — Feeding Behavior; Breast Feeding; Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: Treatment groups: bottle-fed infants
  * Group 1: 10 infants aged 0-4 weeks (+/- 7 days): 0-4 m bottle
  * Group 2: 10 infants aged 4 months (+/- 10 days): 4-6 m bottle
  * Group 3: 10 infants aged 6-10 months (+/- 10 days): 6m+ bottle Control groups: exclusively or prevalently breast-fed infants
  * Group 4: 10 infants aged 0-4 weeks (+/- 7 days)
  * Group 5: 10 infants aged 4 months (+/- 10 days)
  * Group 6: 10 infants aged 6-10 months (+/- 10 days) (at least 2 breastfeeding sessions per day)
  Number of subjects enrolled and allocated: 61 healthy infants, both male and female as follows:
  Treatment groups: bottle-fed infants
  * Group 1: 11 infants aged 0-4 weeks (+/- 7 days): 0-4 m bottle
  * Group 2: 10 infants aged 4 months (+/- 10 days): 4-6 m bottle
  * Group 3: 10 infants aged 6-10 months (+/- 10 days): 6m+ bottle Control groups: exclusively or prevalently breast-fed infants
  * Group 4: 10 infants aged 0-4 weeks (+/- 7 days)
  * Group 5: 10 infants aged 4 months (+/- 10 days)
Masking Description: This was a prospective, open-label, monocentric, interventional clinical study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Feeding Bottle 0m+ (Experimental): 10 infants aged 0-4 weeks (+/- 7 days): 0-4 m bottle. 0-4 months, 250 ml, 2 angled teats: newborn (also referred to as low flow) and infant (also referred to as medium flow), for infants aged 0-4 weeks (+/- 7 days) / over 9 weeks of participation.
  Interventions: Device: infants bottles
- Feeding Bottle 4m+ (Experimental): 10 infants aged 4 months (+/- 10 days): 4-6 m bottle. 4-6 months, 250 ml, non-angled teat), for infants aged 4 months (+/- 10 days) / over 9 weeks of participation.
  Interventions: Device: Infants Bottles
- Feeding Bottle 6m+ (Experimental): 10 infants aged 6-10 months (+/- 10 days): 6m+ bottle. 6 months and over, 250 ml, longer teat) for infants aged form 6 to 10 months (+/- 10 days) / over 9 weeks of participation.
  Interventions: Device: Infants Bottles
- exclusively or prevalently breast-fed infants 0m+ (No Intervention): 10 infants aged 0-4 weeks (+/- 7 days)
- exclusively or prevalently breast-fed infants 4m+ (No Intervention): 10 infants aged 4 months (+/- 10 days)
- exclusively or prevalently breast-fed infants 6m+ (No Intervention): 10 infants aged 6-10 months (+/- 10 days) (at least 2 breastfeeding sessions per day)

INTERVENTIONS:
Device: infants bottles — * angled/inclined teat that remains full of milk throughout the feeding to prevent the risk of air ingestion, gassy colic, hiccups and regurgitation and to keep the infant's neck in the right position;
  * extra-large, soft and rounded base to ensure maximum simulation of the maternal breast and a wide latch on for a correct suckling motion
  * flexors at the base to enhance elasticity and flexibility of the teat
  Other Names: Natural Feeling/Natural Fit 0-4m:
  Arms: Feeding Bottle 0m+
Device: Infants Bottles — * large, rounded and soft teat to ensure maximum simulation of the maternal breast and a wide latch on for a correct suckling motion
  * non-inclined shape of the teat ideal from 4 months onwards, when the colic episodes have subsided and infant has more control of the neck.
  * flexors at the base to enhance elasticity and flexibility of the teat
  Other Names: Natural Feeling/Natural Fit 4-6m:
  Arms: Feeding Bottle 4m+
Device: Infants Bottles — * teat with less rounded base to guarantee tighter lip support, which helps the "sucking" motion.
  * flexors at the base to enhance elasticity and flexibility of the teat
  Other Names: Natural Feeling/Natural Fit 6m+:
  Arms: Feeding Bottle 6m+

SUMMARY:
Breastfeeding is recommended as the ideal form of nutrition for newborns and infants at least for the first 6 months of life by several Institutions such as the American Academy of Pediatrics (AAP) and the World Health Organization (WHO).

When breastfeeding is not possible or not desirable, bottle-feeding, in most cases using a proper infant formula, is the right alternative.

Both facial and cranial growth and development rely on genetic and external stimuli; the latter are provided also by activities of sucking, swallowing and chewing. Considering this, it is important to show the differences between the activities of the muscles (masseter, temporalis and buccinator) in charge of sucking during breastfeeding or bottle-feeding.

The activities of the muscles were evaluated through SLI, which consists of the assessment of muscle functioning by analyzing the displacement of a defined point on a given muscle. This displacement is tracked over time with respect to a fixed frame of reference, thus providing velocity data (i.e. speed) for a certain point on the muscle during muscle contraction. The use of SLI allowed us to determine the activity of oral muscles on the different types of feeding and to compare their strength and activity.

Principal aims of the present study was to assess the activity of the orbicularis oris muscle (OM) and of the masseter, temporalis and buccinator muscles (MM, TM and BM) (i.e. the muscles in charge of sucking during breastfeeding) during breastfeeding and bottle-feeding by means of SLI. The new Chicco feeding bottles Natural Feeling (Natural Fit) 0m+, 4m+ and 6m+ were used according to the age of the infants.

Moreover, the following parameters were evaluated comparing breastfeeding and bottle-feeding: feeding efficiency (measured as ml/minute milk intake considering an interval of 15 minutes) and oxygen saturation during feeding (assessed by pulse oximetry). Moreover colic-like symptoms over 9 weeks (0 to 4 weeks infant only) were evaluated through the Infant Colic Scale.

DETAILED DESCRIPTION:
By means of SLI technique positive preliminary results as regards comparison between bottle feeding with the New Chicco Bottles and breastfeeding were reached; these results allow to conclude that, considering feeding features related to growth and development, bottle-feeding with the new Chicco bottles can biomimic the suction muscular dynamics of breastfeeding.

A proper growth is confirmed in bottle-feeding groups also by means of evaluations of growth parameters, and it is guaranteed by the evaluation of the oxygen saturation during feeding, that is similar among groups.

As regards evaluation of colic underlying causes in infants ages 0-4 weeks it is possible to state that no differences were found in bottle-fed and breastfed infants: given the lack of differences between the groups, whichever the underlying reason for colic symptomatology could exist, it is possible to infer that using one or the other kind of feeding does not have an impact on symptoms, or had a minor one.

As regards the product satisfaction evaluated comparing the bottle-fed groups positive results were reached in all the evaluation, at V2, Week 5 and Week 9, reaching always a mean score > 8.

Notwithstanding the positive results above outlined a confirmatory study, envisaging a bigger sample size, it is advisable, to confirm and emphasize the results already achieved.

For each trial participant the adverse events/serious adverse events occurrences and a brief clinical examination were assessed during Visits. No special or unusual features of the safety evaluations were found.

ELIGIBILITY:
Inclusion Criteria:

* Male and female infants aged 0 to 10 months according to the following:

Group 1: age 0-4 weeks (+/- 7 days) Group 2: age 4 months (+/- 10 days) Group 3: age 6-10 months (+/- 10 days) Group 4: age 0-4 weeks (+/- 7 days) Group 5: age 4 months (+/- 10 days) Group 6: age 6-10 months (+/- 10 days)

* Infants exclusively or prevalently breast- or bottle-fed
* Full-term infants (≥ 37 weeks of gestation) with APGAR at birth (5 min) ≥ 8 by parent report
* Birth weight ≥ 2.5 kg by parent report
* Capability of the parents / legal guardians, according to Investigator's opinion, to fully comprehend the nature of the study
* Parents / legal guardians' written consent to the study and willingness to comply with study procedures

Exclusion Criteria:

* Birth defect, injury or health condition that interferes with sucking, feeding or breathing
* Any medical condition or disease that may affect subject safety or confound study results, including cardiac or neurological defects
* Infants born from twin or multiple pregnancy
* Any other condition that, in the Investigator's opinion, may preclude the subject's ability to safely complete the trial
* Parents / legal guardians uncooperative and/or non-compliant according to Investigator's opinion

Ages: 1 Day to 10 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2014-06-12 (Actual); Primary Completion 2014-10-25 (Actual); Study Completion 2015-01-05 (Actual)

PRIMARY OUTCOMES:
Mean Velocity orbicularis oris (OM) Muscle by means of SLI | Week 2
  To assess the orbicularis oris muscle (OM) and the perioral muscles (masseter, temporalis and buccinator muscles - MM, TM and BM) activity during breast- or bottle-feeding through SLI of the face during a single feeding session considering 3 treatment groups + 3 comparison groups:
  Treatment groups: bottle-fed infants
  * Group 1: age 0-4 weeks (+/- 7 days): 0-4 m bottle
  * Group 2: age 4 months (+/- 10 days): 4-6 m bottle
  * Group 3: age 6-10 months (+/- 10 days): 6m+ bottle Control groups: exclusively or prevalently breast-fed infants
  * Group 4: age 0-4 weeks (+/- 7 days)
  * Group 5: age 4 months (+/- 10 days)
  * Group 6: age 6-10 months (+/- 10 days) (at least 2 breastfeeding sessions per day)
Mean Velocity masseter MM Muscle by means of SLI | week 2
  To assess the orbicularis oris muscle (OM) and the perioral muscles (masseter, temporalis and buccinator muscles - MM, TM and BM) activity during breast- or bottle-feeding through SLI of the face during a single feeding session considering 3 treatment groups + 3 comparison groups:
  Treatment groups: bottle-fed infants
  * Group 1: age 0-4 weeks (+/- 7 days): 0-4 m bottle
  * Group 2: age 4 months (+/- 10 days): 4-6 m bottle
  * Group 3: age 6-10 months (+/- 10 days): 6m+ bottle Control groups: exclusively or prevalently breast-fed infants
  * Group 4: age 0-4 weeks (+/- 7 days)
  * Group 5: age 4 months (+/- 10 days)
  * Group 6: age 6-10 months (+/- 10 days) (at least 2 breastfeeding sessions per day)
Mean Velocity Temporalis Muscle by means of SLI | week 2
  To assess the orbicularis oris muscle (OM) and the perioral muscles (masseter, temporalis and buccinator muscles - MM, TM and BM) activity during breast- or bottle-feeding through SLI of the face during a single feeding session considering 3 treatment groups + 3 comparison groups:
  Treatment groups: bottle-fed infants
  * Group 1: age 0-4 weeks (+/- 7 days): 0-4 m bottle
  * Group 2: age 4 months (+/- 10 days): 4-6 m bottle
  * Group 3: age 6-10 months (+/- 10 days): 6m+ bottle Control groups: exclusively or prevalently breast-fed infants
  * Group 4: age 0-4 weeks (+/- 7 days)
  * Group 5: age 4 months (+/- 10 days)
  * Group 6: age 6-10 months (+/- 10 days) (at least 2 breastfeeding sessions per day)
Mean Velocity Buccinator Muscle by means of SLI | week 2
  To assess the orbicularis oris muscle (OM) and the perioral muscles (masseter, temporalis and buccinator muscles - MM, TM and BM) activity during breast- or bottle-feeding through SLI of the face during a single feeding session considering 3 treatment groups + 3 comparison groups:
  Treatment groups: bottle-fed infants
  * Group 1: age 0-4 weeks (+/- 7 days): 0-4 m bottle
  * Group 2: age 4 months (+/- 10 days): 4-6 m bottle
  * Group 3: age 6-10 months (+/- 10 days): 6m+ bottle Control groups: exclusively or prevalently breast-fed infants
  * Group 4: age 0-4 weeks (+/- 7 days)
  * Group 5: age 4 months (+/- 10 days)
  * Group 6: age 6-10 months (+/- 10 days) (at least 2 breastfeeding sessions per day)

SECONDARY OUTCOMES:
ml/minute milk intake during an interval of 15 minutes | week 2
  To evaluate feeding efficiency (ml/minute milk intake for 15 minutes) during a single feeding session of breast- or bottle-feeding considering each group; week 2;
oxygen saturation | week 2
  To evaluate oxygen saturation through pulse oximetry during a single feeding session of breast- or bottle-feeding considering 3 treatment groups + 3 comparison groups (1, 2, 3, 4, 5, 6); this evaluation was be done at week 2;
infant colic scale | week 5
  To evaluate colic-like symptoms over 9 weeks considering breast- or bottle-feeding groups in 0 to 4 weeks infants only (groups 1 and 4), through the validated Infant Colic Scale at week 5.
  The following items were considered:
  * Cow's milk/soy protein allergy intolerance: Max score 12 Min score 2
  * Immature gastrointestinal system Max score 24 Min score 4
  * Immature central nervous system Max score 48 Min score 8
  * Difficult infant temperament Max score 24 Min score 4
  * Parent infant interaction/Problem infant Max score 24 Min score 4
  * Total score Max score 132 Min score 22 The difference between the study groups were evaluated. The scale was used to evaluate a possible difference between bottle- and breastfed infants, there's no "better" or "worse" outcome. Subscales are summed to compute a total score.
infant colic scale | week9
  To evaluate colic-like symptoms over 9 weeks considering breast- or bottle-feeding groups in 0 to 4 weeks infants only (groups 1 and 4), through the validated Infant Colic Scale at week 9.
  The following items were considered:
  * Cow's milk/soy protein allergy intolerance: Max score 12 Min score 2
  * Immature gastrointestinal system Max score 24 Min score 4
  * Immature central nervous system Max score 48 Min score 8
  * Difficult infant temperament Max score 24 Min score 4
  * Parent infant interaction/Problem infant Max score 24 Min score 4
  * Total score Max score 132 Min score 22 The difference between the study groups were evaluated. The scale was used to evaluate a possible difference between bottle- and breastfed infants, there's no "better" or "worse" outcome. Subscales are summed to compute a total score.
overall product satisfaction (10 points likert scales) | week 2
  Overall product satisfaction at week 2. It is assessed on 0 to 10 points Likert scale; minimum value is 0, maximum is 10, corresponding to minimum and maximum satisfaction. The better outcome corresponds to a score equal to 10.
overall product satisfaction (10 points likert scales) | week 5
  Overall product satisfaction at week 5. It is assessed on 0 to 10 points Likert scale; minimum value is 0, maximum is 10, corresponding to minimum and maximum satisfaction. The better outcome corresponds to a score equal to 10
overall product satisfaction (10 points Likert scales) | week 9
  Overall product satisfaction at week 9. It is assessed on 0 to 10 points Likert scale; minimum value is 0, maximum is 10, corresponding to minimum and maximum satisfaction. The better outcome corresponds to a score equal to 10
Ability of infant to latch onto bottle (10 points Likert scales) | week 2
  Ability of infant to latch onto bottle at week 2. It is assessed on 0 to 10 points Likert scale; minimum value is 0, maximum is 10, corresponding to minimum and maximum satisfaction. The better outcome corresponds to a score equal to 10
Ability of infant to latch onto bottle (10 points Likert scales) | week 5
  Ability of infant to latch onto bottle at week 5
Ability of infant to latch onto bottle (10 points Likert scales) | week 9
  Ability of infant to latch onto bottle at week 9. It is assessed on 0 to 10 points Likert scale; minimum value is 0, maximum is 10, corresponding to minimum and maximum satisfaction. The better outcome corresponds to a score equal to 10
Infant comfort (10 points Likert scales) | week 2
  Infant comfort during feeding at week 2
Infant comfort (10 points Likert scales) | week 5
  Infant comfort during feeding at week 5. It is assessed on 0 to 10 points Likert scale; minimum value is 0, maximum is 10, corresponding to minimum and maximum satisfaction. The better outcome corresponds to a score equal to 10
Infant comfort (10 points Likert scales) | week 9
  Infant comfort during feeding at week 9. It is assessed on 0 to 10 points Likert scale; minimum value is 0, maximum is 10, corresponding to minimum and maximum satisfaction. The better outcome corresponds to a score equal to 10
Ease of use by infant (10 points Likert scales) | week 2
  Ease of use by infant at week 2. It is assessed on 0 to 10 points Likert scale; minimum value is 0, maximum is 10, corresponding to minimum and maximum satisfaction. The better outcome corresponds to a score equal to 10
Immediate acceptance by the infant (10 points Likert scales) | week 2
  Immediate acceptance by the infant at week 2. It is assessed on 0 to 10 points Likert scale; minimum value is 0, maximum is 10, corresponding to minimum and maximum satisfaction. The better outcome corresponds to a score equal to 10